CLINICAL TRIAL: NCT00468416
Title: Evaluation of NiTi Shape Memory End-to-End Compression Anastomosis Ring (CAR) for Compression Anastomosis in Anterior Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rabin Medical Center (Other); Kaplan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-43-01-2
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Compression Anastomosis Ring (CAR)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the NiTi CAR device in the creation of colorectal anastomosis

ELIGIBILITY:
Inclusion Criteria:

* Patient age over 18 years
* Patient scheduled for colorectal cancer surgery
* Patient is able to comprehend and sign the Informed Consent Form

Exclusion Criteria:

* Patient has known allergy to nickel
* Patient with bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection
* Patients who are participating in another trial
* Patient on regular steroid medication
* Patients who are undergoing a stoma
* Patients with contraindications to general anesthesia
* Patient with preexisting sphincter problems or evidence of extensive local disease in the pelvis
* Patients after radiation
* Patients who refuse consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-02; Study Completion 2008-02

PRIMARY OUTCOMES:
Functioning anastomosis and no occurrence of adverse events related to device use | During hospitalization and one month post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Tulchinsky, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel